CLINICAL TRIAL: NCT06737744
Title: Active Games for Increasing Social and Emotional Competencies of Young Adults in Probation System: a One-Sample Trial Study in Izmir City in Turkiye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Inci Derya YUCEL, Lecturer, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC.20.16.1; 604730EPP120181UKEPPKA3IPISOC- (Other Grant/Funding Number: European Commission Erasmus+ Programme)
Record Dates: First submitted 2024-11-28; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Substance Use Disorder; Sports; Competency Based Education; Psychological Well Being; Addiction
Keywords: substance use disorder; physical activity; youth justice; probation service; education; mental health well being; addiction
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being; Behavior, Addictive; Motor Activity

STUDY DESIGN:
Intervention Model Description: The recruitment of this study was conducted in accordance with a pre-established plan, which entailed the selection of a total of 50 participants who met the established inclusion and exclusion criteria. These participants were divided into groups of 7-10 individuals. Each participant was required to attend a minimum of 2 and a maximum of 4 different sessions. In each session, the participants were exposed to games with varying levels of difficulty and content, which were designed to develop the specified competencies and skills outlined in the CASEL model at different levels. The majority of these games were group games that involved low or moderate physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AG4C intervention group (Experimental)
  Interventions: Other: Active Games for Change (AG4C); Behavioral: Active Games for Change Group Working

INTERVENTIONS:
Other: Active Games for Change (AG4C) — This intervention was carried out in Turkiye within the Erasmus+ Key Action 3 project titled Active Games for Change (AG4C). The programme included a series of innovative, face-to-face active games with a non-formal approach that prioritised physical activity, specifically designed to support the development of social and emotional competencies identified for the first time in the field in a probation directorate serving young adult offenders.
Behavioral: Active Games for Change Group Working — The Active Games for Change intervention program was implemented in Izmir, Türkiye within the Erasmus+ Key Action 3 project titled Active Games for Change (AG4C). The AG4C intervention program included a series of innovative, face-to-face active games with a non-formal approach that prioritised support for developing social and emotional competencies of young adults with substance use problems, for the first time in the field.
  Other Names: "Active Games for Change; AG4C

SUMMARY:
Objective: The goal of this one-sample clinical trial is to implement active games, including physical activities, that support the social and emotional competencies of individuals in probation sentence.

Methods: The study was carried out with 50 young adult offenders. The Collaborative for Academic, Social, and Emotional Learning (CASEL) model, which defines five social and emotional skills (self-awareness, self-management, responsible decision making, relationship skills, social awareness), was used to support observation and game design. The present study involved the codesign of a total of 18 active games to develop these five competencies. The primary outcomes of the research were increased mental well-being and increased social emotional skills in participants receiving the AG4C program. The secondary outcome of the research was the regular participation of the participants in the program. In this study, two hypotheses were tested: "The ActiveGames4Change programme increases the psychological wellbeing of young adults on probation" and "The ActiveGames4Change programme increases the 5 basic skills of young adults on probation. This study was carried out with 50 young adult offender individuals (48 male and 2 female) who received probation measures in accordance with the court or prosecutor's decision for different crimes. The CASEL model, which defines social and emotional skills, was used to support observation and game design because it determines the characteristics of young people who are in the execution process. The skill set proposed by the CASEL model included skills such as "self-awareness", "self-management", "social awareness", "relationship skills" and "responsible decision-making".

The Wilcoxon signed-rank test was employed to examine the impact of the intervention on participants' progression of competency levels before and after the intervention.

DETAILED DESCRIPTION:
This work involved the codesign of 18 active games to develop five core competencies. Each game was designed with three levels: Level 1 games require less complex social and emotional competencies; Level 2 acts as a bridge to cement and develop those established in Level 1; and Level 3 requires either more competencies or competencies used at a higher level of difficulty. Nine of them were applied to 38 participants during 4 sessions at different times in the present study between 14/12/2021 and 09/02/2022.

Nine of the 18 games could not be played due to the limitations of the COVID-19 pandemic. It was carried out by 10 trainers with 50 (including 12 dropouts) young individuals at the Izmir Probation Directorate in Turkiye. Since the current physical conditions of the institution were not suitable, a full-fledged sports hall affiliated with the municipality was implemented as a result of cooperation with a local governmental institution. The Turkish version of the Warwick-Edinburgh Well-being Scale (WEMWBS) was used by the participants before and at the end of the AG4C Program, which evaluated the five SECs mentioned above. All measurements were obtained by asking the participant by the instructor/educator or researcher instead of self-reporting.

Thus, the biases caused by the participants were minimized by ensuring that the participants perceived the questions correctly.

Eighteen games were designed within the CASEL framework, and each game had three levels, which means that there were six games at each level. The game cards were developed, which included instructions about how to implement the game for educators and learners (probationers). All games were also available on the specially designed AG4C App (www.activegames4change.org/ag4c-app.html), where progress data could also be captured.

After the games were designed, 10 educators in a probation service were trained by two master trainers to enable them to test the games program with young people as well as to gather both pre- and post-intervention data. Additionally, the educators (n=10) conducted evaluations of the games that they had implemented for the participants.

A comprehensive training package was provided to the educators of the Izmir Probation Directorate. The package consisted of 18 games and online theoretical and practical training with video tutorials. The games were collaboratively developed in English by experts through expert panels and 2 validation workshops, all of which involved AG4C project partners, before they were adapted for usage. Subsequently, the researcher translated all the materials from English into Turkish in preparation for use in the pilot program in Turkiye.

ELIGIBILITY:
Inclusion Criteria:

* being between 18 and 30 years old
* having any kind of criminal background under probation supervision
* having at least four months left on their probation sentence.

Exclusion Criteria:

* having physical health issues
* severe mental disorders such as schizophrenia, borderline personality disorder, and antisocial personality disorder.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
The total score of the mental well-being | From enrollment to the end of intervention at 8 weeks
  The total score for mental well-being was obtained from the Warwick Edinburgh Mental Well-being Scale (WEMWBS) in Turkish, completed by participants verbally with the assistance of educators, before and at the end of the "Active Games 4 Change" intervention. WEMWBS was developed and validated for multicultural use and is available in Turkish. The scale consists of 14 positive items and has a 5-point Likert-type answer key. The lowest score is 14 points and the highest score is 70 points. High scores obtained from the scale indicate high mental (psychological) well-being. The Turkish version of WEMWBS retains the single-factor structure of the original scale and demonstrates robust validity and reliability. The queries were cross-referenced with CASEL's core social-emotional competencies to ensure each was covered by at least one question.
Social Emotional Skills | From enrollment to the end of intervention at 8 weeks
  Collaborative for Academic, Social and Emotional Learning(CASEL) defines 5 social emotional skills:Self-Awareness(SA1), Social Awareness(SA2), Self-Management(SM) Relationship skills(R) and Responsible Decision-making(RD) which guided the design of 18 games to develop these skills.To observe the five CASEL social emotional skills of the participants,Warwick-Edinburgh Well-being Scale (WEMWBS) items were evaluated, and the team of this research determined which items best described each skill.The queries WEMWBS were cross-referenced with CASEL's skills to ensure each was covered by at least one item in WEMWBS.A matching process aligned CASEL skills with WEMWBS scoring,generating sub-scores to assess each skill's progress.Higher scores indicated greater progress.The matched items with points:SA1-items 2,3,8,10(min:4,max:20);SA2-item 4(min:1,max:5);SM-items 1,5,13(min:3,max:15);R-items 9,12(min:2,max:10);RD-items 6,7,11(min:3,max:15).Each response was scored on a scale of 1 to 5 points.

SECONDARY OUTCOMES:
Regular participation of the participants in the program | From enrollment to the end of intervention at 8 weeks
  Regular participation is defined as attending at least 2 out of 4 sessions during the 8-week intervention. Participation rates were recorded by educators using a participant registration form which was created by the researcher team.
  Unit of Measure: Percentage of participants meeting the attendance criteria (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Institute on Drug Abuse, Toxicology and Pharmaceutical Science, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wigelsworth M. SPECTRUM': Social, psychological, emotional, concepts of self, and resilience: Understanding and measurement. 2017
- [Background] Keldal G. Warwick-Edinburgh Turkish Version of the Warwick-Edinburgh Mental Well-Being Scale: A validity and reliability study. The Journal of Happiness & Well-Being. 2015; 3(1), 103-115.
- [Background] WHO Guidelines on Physical Activity and Sedentary Behaviour. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK566045/ PMID 33369898
- [Background] Moyles, J. EBOOK: The Excellence of Play. McGraw-Hill Education (UK). 2014
- [Derived] Yucel ID, Yararbas G. Active games for increasing social and emotional competencies of young adults in probation system: a one-sample trial study in Izmir city in Turkiye. BMC Psychol. 2024 Dec 31;12(1):797. doi: 10.1186/s40359-024-02309-0. PMID 39741356
- See also: Leading Change Through Activity & Sports - A Handbook for Leaders about the AG4C Methodology — http://www.activegames4change.org/uploads/9/7/7/2/97721820/leading_change_through_activity___sports_%E2%80%93_a_handbook_for_leaders_about_the_ag4c_methodology.pdf#page=17.57